CLINICAL TRIAL: NCT04195347
Title: CRSPA: Phase I/II Study of CM4620 to Reduce the Severity of Pancreatitis Due to Asparaginase
Brief Title: Study of CM4620 to Reduce the Severity of Pancreatitis Due to Asparaginase
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: CalciMedica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRSPA; NCI-2019-08205 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2019-11-25; First posted 2019-12-11 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Acute Pancreatitis
Keywords: Acute Pancreatitis; Asparaginase; Asparaginase Associated Pancreatitis; Acute Lymphoblastic Leukemia; Acute Lymphoblastic Lymphoma; CM4620; Children; SIRS; Systemic Inflammatory Response; Young Adults
MeSH Terms: conditions — Pancreatitis; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — zegocractin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CM4620 Treatment (Experimental): Phase I:
  Cohort 1 patients receive CM4620 IV at dose level 1 on days 1-4. Cohort 2 patients receive CM4620 IV at dose level 2 on days 1-4. Cohort 3 patients receive CM4620 IV at either dose level 1 or 2 on days 1-4
  Phase II:
  Patients will receive CM4620 IV on days 1-4 at the recommended Phase II dose (RP2D) as determined in Phase I.
  Interventions: Drug: CM4620

INTERVENTIONS:
Drug: CM4620 — IV
  Other Names: CM4620-IE

SUMMARY:
This is a phase I/II clinical trial assessing the tolerability and efficacy of CM4620 in children and young adults with acute pancreatitis caused by asparaginase. The tolerability of CM4620 when given to patients receiving frontline chemotherapy will be determined. The effectiveness in reducing the severity of pancreatitis will be estimated.

Primary Objectives

To assess the safety of CM4620 administration in children and young adults with asparaginase associated pancreatitis (AAP).

To profile dose-limiting toxicities and responses of the patients treated in the dose-finding phase.

To estimate the efficacy of CM4620 to prevent pseudocyst or necrotizing pancreatitis in children with AAP.

Secondary Objectives

To determine the effect of CM4620 on the incidence of severe pancreatitis

To determine the effect of CM4620 on the incidence of Systemic Inflammatory Response Syndrome (SIRS).

DETAILED DESCRIPTION:
This is an open label safety and efficacy evaluation with comparison of toxicity to a historical control population (TOTXVI). There will be 3 cohorts of patients enrolled, and the dose for each cohort will be determined based on the toxicities experienced in the ongoing and prior cohorts.

An initial 9 patients (cohort 1) will be enrolled and will receive dose level 1 and monitored for toxicity. If the therapy is well tolerated, 6 patients (cohort 2) will be treated at dose level 2. Subsequent enrollment of 9 patients (cohort 3) will be at either dose level 1 or 2 based on tolerability. The keyboard design will be used to determine the dosing for cohorts 2 and 3. Additional patients will be enrolled at the recommended phase II dose (RP2D) until a total of 24 patients have been treated at that dose, including any treated during the dose-finding phase.

CM4620 will be given days 1-4 as an IV infusion beginning within 36 hours of the onset of acute pancreatitis associated abdominal pain and within 8 hours of enrollment. For patients with prior abdominal pain or in those unable to communicate the location/characteristic of their pain, a change in the characteristic of the pain or new enzyme elevation/imaging findings after previously normal studies will determine the timing of onset of pancreatitis.

Patients will be followed for about 4 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Acute pancreatitis with elevation of amylase OR lipase ≥ 3x the upper limit of normal AND at least 1 of: abdominal pain consistent with acute pancreatitis OR imaging findings consistent with acute pancreatitis.
* Receipt of any form of asparaginase within the prior 49 days.
* Patient with acute lymphoblastic leukemia/ lymphoma age < 22 years receiving therapy with curative intent.

Exclusion Criteria:

* Prior episode of pancreatitis.
* QTc at baseline > 450 msec.
* Creatinine > 3x the upper limit of normal for age or total bilirubin >3x the upper limit for normal for age without evidence of leukemic infiltrate or hemolysis.
* Receipt of another investigational agent within the prior 7 days.
* History of allergy to eggs or known hypersensitivity to any component of CM4620.
* Positive pregnancy test or breastfeeding. Females of childbearing potential must have a negative urine or serum pregnancy test prior to enrollment. Males and females of childbearing potential must agree to use effective contraception for at least twelve months following the completion of therapy.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
The number of CTCAE grade 3-5 events | Within 28 days of receiving the medication
  Drug safety measuring the number of CTCAE grade 3-5 events
Responses to CM4620 | 28-35 days after study entry.
  We will evaluate the rate of pancreatic necrosis or pseudocyst formation using radiographic imaging

SECONDARY OUTCOMES:
Effect of CM4620 measured by levels of pancreatic enzymes | 72 hours after study entry
  Pancreatitis measured by levels of pancreatic enzymes
Effect of CM4620: Necrosis | 28-35 days from study entry
  Necrosis measured by levels of pancreatic enzymes
Effect of CM4620: Pseudocyst | 28-35 days from study entry
  Pseudocyst measured by levels of pancreatic enzymes
Effect of CM4620: Incidence of SIRS | 48-72 hours after study entry
  Presence or absence of systemic inflammatory response syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Seth E. Karol, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - Novant Health Presbyterian Hemby Children's Hospital, Charlotte, North Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: ClinicalTrials Open at St. Jude — http://www.stjude.org/protocols